CLINICAL TRIAL: NCT04996537
Title: Nantou Hospital, Ministry of Health and Welfare
Brief Title: Effectiveness of Flipped Learning on Nurses' Knowledge, Attitude, and Self-efficacy in Pressure Injury Prevention
Acronym: KAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wen-Yi Chao (Other Government)
Responsible Party: Sponsor-Investigator, Wen-Yi Chao, Principal Investigator, Nantou Hospital
Organization: Nantou Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nantou Hospital
Record Dates: First submitted 2021-07-22; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Educational Problems
Keywords: knowledge; attitude; self-efficacy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Quasi-experimental research, with repeated measures research design
Who Masked: Participant
Masking Description: Both the experimental group and the control group received the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-video with pressure injury(PI) education (Experimental): The experimental group's flipped education and training courses adopt a digital learning method and provide a digital learning platform. Log in according to personal account and password, and learn the curriculum units planned by the researcher in order: "Prevention and management of stressful injury care" as the main axis, enter the digital platform The provided video audio-visual digital teaching materials, combined with clinical situational learning, are equipped with basic knowledge learning, in-class test questions, and unit review, and can open courses for self-study anytime and anywhere, regardless of time and space constraints.
  Interventions: Other: Micro-video digiral learning
- NIS with PI education (Active Comparator): At the login interface of the Nursing Information System (NIS) used by the nursing staff daily, a link to the lecture notes (PDF file) of the course on prevention of stress injury is attached, and the nursing staff can view or download them according to their needs. Learn. At the same time, it provides a digital learning platform to download the self-study course handouts (PDF files) and complete the basic demography, pre-test, and post-test data on the platform.
  Interventions: Other: Micro-video digiral learning

INTERVENTIONS:
Other: Micro-video digiral learning — On the digital platform, you can accept courses anytime, anywhere, and repeat learning, answering, leaving messages, or interacting with lecturers.
  Other Names: digital platform learning

SUMMARY:
The occurrence of pressure injuries mainly comes from disabled patients who are bedridden for a long time. According to a report from the Ministry of Health and Welfare, about one-tenth of chronic patients need to be bedridden for a long time, and pressure injuries account for the most in the comorbidities of bedridden for a long time. The main cause of pressure injury is the natural aging of the patient's body and long-term bed rest so that it is difficult to detect physical stress and cannot change the posture within an effective time to reduce the pressure, which is prone to pressure injury. The prevalence rates of stress injuries in various countries are 13-23% in the Netherlands, 10-15% in the United States, and 8-23% in Europe. In addition, studies have also shown that the prevalence of stress injuries in the elderly in the UK is 0.31-0.70%. The incidence rate is 0.18-3.36% and these two indicators are increasing year by year; in Taiwan, related surveys show that the prevalence rate of pressure injury in hospitalized patients is 7.53%, and the incidence rate of pressure injury in bedridden patients is 36.8%. According to a National Pressure Ulcer Advisory Panel (NPUAP) survey, the prevalence rate of stress injuries in acute wards ranges from 0.1% to 17%, and the incidence rate is 0.4% to 38%. The prevalence of intensive care units The prevalence rate is higher than 41%, the incidence rate is higher than 33%, the prevalence rate of long-term care is 2.3% -28%, the prevalence rate is 2.2%-23.9%, the prevalence rate of nursing homes is 0% -29%, and the prevalence rate is 0%- 17%. In addition, NPUAP estimates in 1989 show that the average medical cost for each stress injury case ranges from 2,000 to 30,000 US dollars, while the medical cost for each stress injury patient in Taiwan is about NT 7,000 to 80,000. If the knowledge of stress injury prevention can be improved, the number of outpatient visits will be reduced, and the occurrence of stress injury will also be reduced. In summary, under the trend of aging development, stress injury management and care are important issues of medical quality.

DETAILED DESCRIPTION:
The purpose of this research is to integrate the past education that affects nursing staff to receive care for stress injuries and to explore the intervention of different education measures, including conventional education methods and digital flipped education methods, to measure nursing staff Effectiveness in learning about the knowledge, attitude, self-awareness and self-efficacy of pressure injury management.

ELIGIBILITY:
Inclusion Criteria:

1. Full-time or part-time nursing staff registered in the research site and engaged in front-line clinical care or nursing-related administrative services;
2. Those who agree to participate in the research and provide informed consent.

Exclusion Criteria:

Nursing student

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-16 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
knowledge | 20minutes
  This tool can be used to assess medical staff's knowledge of stress injury prevention. Developed by Pieper and Mott in 1995 (Reference: Pieper B, Mott M. Nurses' knowledge of pressure ulcer prevention, staging, and description. Adv Wound Care 1995; 8: 34-48.)
Attitude | 3-5minutes
  Moore and Price (2004) researched to develop tools to evaluate nurses' attitudes towards pressure ulcer prevention. The tool includes 11 items, which are scored according to the Likert scale five-point scale, from 5 (strongly disagree) to 1 (strongly agree)
self- efficacy | 3-5minutes
  PUM-SES aims to evaluate the self-efficacy of nursing staff in managing stress injuries and was published in 2019 (Dellafiore et al., 2019). There are 10 items in the PUM-SES scale, including four areas: evaluation, planning, supervision, and decision-making.

IPD SHARING:
Plan to Share IPD: No